CLINICAL TRIAL: NCT02126826
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1026706 in Male and Female Healthy Subjects and Patients With Osteoarthritis of the Knee (Randomised, Double-blind, Placebo-controlled Within the Dose Groups, Clinical Phase I)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1026706 in Male and Female Healthy Subjects and Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.2; 2012-005690-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (2):
- Placebo to BI 1026706 (Placebo Comparator): Multiple Rising Doses Placebo to BI 1026706
  Interventions: Drug: Placebo to BI 1026706
- BI 1026706 (Experimental): Multiple Rising Doses BI 1026706
  Interventions: Drug: BI 1026706

INTERVENTIONS:
Drug: BI 1026706 — Multiple Rising Doses (oral solution, tablet)
  Arms: BI 1026706
Drug: Placebo to BI 1026706 — Multiple Rising Doses (oral solution / tablet, identical to active treatment)
  Arms: Placebo to BI 1026706

SUMMARY:
* To investigate the safety and tolerability of BI 1026706 in male and female healthy subjects and osteoarthritis (OA) patients following oral administration of repeated rising doses
* To explore the pharmacokinetics after multiple rising doses of BI 1026706 in male and female healthy subjects and OA patients
* The assessment of pharmacodynamics in OA patients

ELIGIBILITY:
Inclusion criteria:

1. Males or females without any clinically relevant medical disorders according to the investigator's assessment, as based on the following: a complete medical history including a physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, and clinical laboratory tests
2. For OA patients: Evidence of OA of the knee by radiography or by magnetic resonance tomography (Kellgren-Lawrence grade 1, 2, or 3; excluding grades 0 and 4) of the knee (tibiofemoral joint only) within the last 5 years consistent with the clinical diagnosis of osteoarthritis of the knee according to American College of Rheumatology (ACR) guidelines
3. For OA patients: American Rheumatism Association (ARA) functional class I, II, or III
4. For OA patients: Average pain in the index knee over the previous 48 hours greater than or equal to 4 on the 11-item Likert scale at two time points: 1) at screening (if not on analgesic medication) or after 3 days of wash-out of analgesic medication, and 2) in the evening prior to randomisation
5. For OA patients: Presence of bothersome OA related pain for most days within the last month prior to screening at the investigator's discretion, or pain requiring analgesic treatment on more than 3 days per week during the last month prior to screening.
6. Age 35 to 65 years (inclusive)
7. BMI (Body Mass Index) 18.5 to 33 kg/m2 (inclusive)
8. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
9. Females who meet any of the following criteria from at least 30 days before the first study drug administration and until 30 days after trial completion:

   * using adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral contraceptives, intrauterine device (IUD)
   * sexually abstinent
   * have a vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
   * surgically sterilised (including hysterectomy)
   * postmenopausal defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of FSH (Follicle Stimulating Hormon) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion criteria:

1. Any finding in the medical examination (including Blood Pressure, Pulse Rate or electrocardiogram) deviating from normal and judged clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug(s)
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1320.2.2 Boehringer Ingelheim Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo HV: Healthy volunteers (HV) received a matching placebo containing quinine sulphate dehydrate, once daily for 12 days.
- 50mg BI 1026706 HV: Healthy volunteers (HV) received 50mg BI 1026706 once daily on days 1 to 12 in the form of a powder for oral solution.
- 100mg BI 1026706 HV: Healthy volunteers (HV) received 100mg BI 1026706 once daily on days 1 to 12 in the form of a powder for oral solution.
- 300mg BI 1026706 HV: Healthy volunteers (HV) received 300mg BI 1026706 once daily on days 1 to 12 in the form of a powder for oral solution.
- Placebo OA: Patients with osteoarthritis (OA) received a matching placebo containing quinine sulphate dehydrate, once daily for 12 days.
- 200mg BI 1026706 OA: Patients with osteoarthritis received 200mg BI 1026706 once daily on days 1 to 12 in the form of a powder for oral solution.
- 100mg BI 1026706 BID OA: Patients with osteoarthritis received oral administration of 100mg BI 1026706 tablets twice daily (BID) on days 2 to 11 and once daily on days 1 and 12.
Period: Overall Study
Arm/Group | Placebo HV | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | Placebo OA | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Started | 9 | 9 | 9 | 9 | 5 | 9 | 8
Completed | 9 | 9 | 9 | 8 | 5 | 9 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) which included all randomised patients and healthy subjects who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo HV | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | Placebo OA | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 5 | 9 | 8 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (9.6) | 43.6 (5.3) | 50.1 (11.8) | 48.7 (8.8) | 50.2 (10.8) | 49.8 (8.4) | 58.1 (4.9) | 49.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 4 | 3 | 2 | 5 | 28
  Male | 3 | 5 | 5 | 5 | 2 | 7 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug Related Adverse Events
Description: Percentage of subjects with drug related adverse events (AEs)
Time Frame: From first drug administration until 3 days after last drug administration, 15 days
Population: Treated set (TS)
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo HV | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | Placebo OA | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 5 | 9 | 8
Percentage of participants | 22.2 | 22.2 | 11.1 | 66.7 | 60.0 | 55.6 | 37.5

2. Secondary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax)
Time Frame: 1 hour (h) 30 minutes (min) before first drug admin and 10min, 20min, 30min, 45min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 14h and 23h 55min after first drug admin
Population: Pharmacokinetic set (PKS) which included all patients and healthy subjects in the TS who provided at least 1 PK endpoint value without relevant protocol deviations with respect to the evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
nmol/L | 423 (31.2) | 1010 (25.3) | 1600 (54.3) | 1730 (36.1) | 578 (53.6)
Statistical Analysis 1: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 300mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 300mg; Test type: Superiority or Other; ANCOVA; Slope = 0.7865, 90% CI 2-sided [0.6193 to 0.9537]
Statistical Analysis 2: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 200mg; Test type: Superiority or Other; ANCOVA; Slope = 1.0171, 90% CI 2-sided [0.8378 to 1.1964]

3. Secondary Outcome: Time From Dosing to Maximum Measured Concentration (Tmax)
Description: Time from dosing to maximum measured concentration of the analyte in plasma (Tmax)
Time Frame: as for outcome 2
Population: PKS
Measure: Median (Full Range); unit: hours
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
hours | 0.52 [0.47 to 2.00] | 0.52 [0.33 to 0.98] | 0.69 [0.37 to 2.53] | 0.75 [0.50 to 1.08] | 1.53 [0.75 to 8.13]

4. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Interval From 0 Extrapolated to 24h (AUC0-24)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 24 hours (h) (AUC0-24).
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
nmol*h/L | 1230 (44.9) | 2790 (26.7) | 6410 (66.2) | 5530 (44.9) | 2790 (58.5)
Statistical Analysis 1: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 300mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 300mg; Test type: Superiority or Other; ANCOVA; Slope = 0.9511, 90% CI 2-sided [0.7654 to 1.1367]
Statistical Analysis 2: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 200mg; Test type: Superiority or Other; ANCOVA; Slope = 1.0834, 90% CI 2-sided [0.8655 to 1.3013]

5. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Interval From 0 Extrapolated to 12h (AUC0-12)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to 12 hours (h) (AUC0-12).
Time Frame: 1 hour (h) 30 minutes (min) before first drug admin and 10min, 20min, 30min, 45min, 1h, 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h and 12h after first drug admin
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
nmol*h/L | 1050 (41.3) | 2370 (27.8) | 5080 (63.6) | 4720 (45.1) | 2290 (54.2)

6. Secondary Outcome: Maximum Measured Concentration at Steady-state (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady-state over a uniform dosing interval τ (Cmax,ss).
Time Frame: 5 minutes (min) before drug admin on day 12 and 10min, 20min, 30min, 45min, 1 hour (h), 1h 30min, 2h, 2h 30min, 3h, 4h, 6h, 8h, 10h, 12h, 14h and 24h after drug admin on day 12
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
nmol/L | 485 (37.4) | 1190 (26.1) | 1800 (43.3) | 2040 (27.0) | 723 (65.1)
Statistical Analysis 1: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 300mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 300mg; Test type: Superiority or Other; ANCOVA; Slope = 0.7832, 90% CI 2-sided [0.6235 to 0.9428]
Statistical Analysis 2: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 200mg; Test type: Superiority or Other; ANCOVA; Slope = 1.0365, 90% CI 2-sided [0.8593 to 1.2137]

7. Secondary Outcome: Time From Last Dosing to Maximum Measured Concentration at Steady-state (Tmax,ss)
Description: Time from last dosing to maximum concentration of the analyte in plasma at steady-state (Tmax,ss).
Time Frame: as for outcome 6
Population: PKS
Measure: Median (Full Range); unit: hours
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
hours | 0.53 [0.30 to 1.00] | 0.52 [0.35 to 1.02] | 0.58 [0.45 to 1.02] | 0.58 [0.33 to 1.05] | 1.13 [0.73 to 3.03]

8. Secondary Outcome: Area Under the Concentration-time Curve at Steady-state (AUCτ,ss)
Description: Area under the concentration-time curve of the analyte in plasma at steady-state over a uniform dosing interval τ (AUCτ,ss).
Time Frame: as for outcome 6
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8
nmol*h/L | 1610 (51.4) | 4080 (24.5) | 8550 (44.5) | 7200 (38.9) | 3280 (61.3)
Statistical Analysis 1: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 300mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 300mg; Test type: Superiority or Other; ANCOVA; Slope = 0.9433, 90% CI 2-sided [0.7744 to 1.1122]
Statistical Analysis 2: Comparison: 50mg BI 1026706 HV vs 100mg BI 1026706 HV vs 200mg BI 1026706 OA; Investigation of dose proportionality - dose groups 50mg to 200mg; Test type: Superiority or Other; ANCOVA; Slope = 1.0810, 90% CI 2-sided [0.8583 to 1.3037]

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 days after last drug administration, 15 days
Arm/Group | Placebo HV | 50mg BI 1026706 HV | 100mg BI 1026706 HV | 300mg BI 1026706 HV | Placebo OA | 200mg BI 1026706 OA | 100mg BI 1026706 BID OA
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/5 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 5/9 | 3/9 | 2/9 | 6/9 | 3/5 | 6/9 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo HV (N=9) | 50mg BI 1026706 HV (N=9) | 100mg BI 1026706 HV (N=9) | 300mg BI 1026706 HV (N=9) | Placebo OA (N=5) | 200mg BI 1026706 OA (N=9) | 100mg BI 1026706 BID OA (N=8)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 3 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.